CLINICAL TRIAL: NCT06921850
Title: A Multicenter, Open-Label Study to Assess The Pharmacokinetics And Safety of Bimekizumab in Pubertal Children And Adolescents With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Bimekizumab in Children and Adolescents With Moderate to Severe Hidradenitis Suppurativa
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS0006; 2023-505323-31 (Registry Identifier: EU Clinical Trials); U1111-1316-5308 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Bimekizumab; HS; Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bimekizumab (Experimental): Study participants will receive a bimekizumab dose which is weight-dependent.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab will be administered at pre-specified timepoints.

SUMMARY:
The purpose of the study is to assess the PK of bimekizumab following subcutaneous (sc) administration in study participants with moderate to severe hidradenitis suppurativa (HS)

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 12 to <18 years of age at the time of informed consent/assent, at Tanner stage 2 or more, for the first 8 participants only, followed by also including participants ≥9 to <18 years of age at Tanner stage 2 or more.
* Study participant must have a diagnosis of HS for at least 6 months prior to the Baseline Visit.
* Study participant must have moderate to severe HS, defined as a total of ≥5 inflammatory lesions (ie, the sum of abscesses and inflammatory nodules), as assessed at both the Screening and Baseline Visits.
* Study participant must have HS lesions present in at least 2 distinct anatomic areas, 1 of which must be at least Hurley Stage II or III, as assessed at both the Screening and Baseline Visits.
* Study participant must have had a history of inadequate response to a course of a systemic antibiotic for treatment of HS
* Study participant must weigh ≥30kg at the Screening Visit.

Exclusion Criteria:

* Study participant has a draining tunnel count of >20 at either the Screening or Baseline Visits.
* Study participant has experienced primary failure (no response within 12 weeks) to 1 or more IL 17 biologic response modifiers (eg, brodalumab, ixekizumab, secukinumab) OR primary failure to more than 1 biologic response modifier other than an IL-17 biologic response modifier.
* Study participant has previously participated in this study or has received previous therapy with bimekizumab.
* Study participant has a history of IBD or symptoms suggestive of IBD.
* History of active tuberculosis unless successfully treated, latent TB unless prophylactically treated
* Study participant has an active infection or history of infections (such as serious infection, chronic infections, opportunistic infections, unusually severe infections)
* Study participant has received drugs outside the specified timeframes relative to the Baseline Visit or receives prohibited concomitant treatments
* Study participant has the presence of active suicidal ideation, or positive suicide behavior,
* Study participant diagnosed with severe depression in the past 6 months prior to the Screening Visit.
* Study participant has a history of psychiatric inpatient hospitalization within the past year before enrolling into the study.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Plasma bimekizumab concentrations at Week 16 | At Week 16
  Plasma samples will be collected prior to dosing for measurement of plasma concentrations of bimekizumab at the specified timepoint.

SECONDARY OUTCOMES:
Exposure-adjusted incidence rate of Treatment- Emergent Adverse Events (TEAEs) during the Initial Treatment Period | From Baseline until end of the Initial Treatment Period (up to 16 weeks)
  The TEAEs adjusted by duration of exposure to study treatment are scaled such that it provides an incidence rate per 100 patient-years. If a participant has multiple events, the time of exposure will be calculated to first occurrence of the AE being considered. If a participant has no events, the total time at risk will be used. An Adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to IMP.
Exposure-adjusted incidence rate of Serious TEAEs during the Initial Treatment Period | From Baseline until end of the Initial Treatment Period (up to 16 weeks)
  The TEAEs adjusted by duration of exposure to study treatment are scaled such that it provides an incidence rate per 100 patient-years. If a participant has multiple events, the time of exposure will be calculated to first occurrence of the AE being considered. If a participant has no events, the total time at risk will be used. A SAE is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events
Exposure-adjusted incidence rate of TEAEs leading to withdrawal during the Initial Treatment Period | From Baseline until end of the Initial Treatment Period (up to 16 weeks)
  The TEAEs adjusted by duration of exposure to study treatment are scaled such that it provides an incidence rate per 100 patient-years. If a participant has multiple events, the time of exposure will be calculated to first occurrence of the AE being considered. If a participant has no events, the total time at risk will be used. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to IMP.
Exposure-adjusted incidence rate of Selected Safety Topics of Interest (including incidence of infections [serious, opportunistic, fungal, and TB], IBD, and injection site reactions) over the Initial Treatment Period | Up to Week 16
  Safety topics of interest for this study include events for which special monitoring will be for infections (serious, opportunistic, fungal, and tuberculosis [TB]), inflammatory bowel disease (IBD), and injection site reactions.
Mean Change from Baseline in vital signs (Systolic Blood Pressure and Diastolic Blood Pressure) at Week 16 | Baseline and Week 16
  Blood pressure (Systolic Blood Pressure and Diastolic Blood Pressure) will be measured in millimeters of mercury (mmHg).
Mean Change from Baseline in vital sign (Pulse rate) at Week 16 | Baseline and Week 16
  Pulse Rate will be measured in beats per minute (beats/min).
Mean Change from Baseline in Biochemistry Laboratory Analyses (glucose, potassium, sodium, calcium) at Weeks 4,12, and 16 | Baseline, Weeks 4, 12, and 16
  Glucose, potassium, sodium and calcium will be measured in millimoles per liter (mmol/L).
Mean Change from Baseline in Biochemistry Laboratory Analyses (total bilirubin and direct bilirubin, total protein, blood urea nitrogen, and creatinine) at Weeks 4,12, and 16 | Baseline, Weeks 4, 12, and 16
  Biochemistry parameters (total bilirubin and direct bilirubin, total protein, blood urea nitrogen [BUN], and creatinine) will be measured in micromols per liter (μmol/L).
Mean Change from Baseline in Biochemistry Laboratory Analyses (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase) at Weeks 4,12, and 16 | Baseline, Weeks 4, 12, and 16
  Biochemistry parameters (alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT) will be measured in units per liter (U/L).
Mean Change from Baseline in Hematology Laboratory Analyses (hemoglobin) at Weeks 4,12, and 16 | Baseline, Weeks 4, 12, and 16
  Hemoglobin will be measured in grams per liter (g/L).
Mean Change from Baseline in Hematology Laboratory Analyses (hematocrit) at Weeks 4,12, and 16 | Baseline, Weeks 4, 12, and 16
  Hematocrit will be measured in volume percentage (%) of red blood cells in blood.
Mean Change from Baseline in Hematology Laboratory Analyses (platelets, leukocytes, neutrophils, lymphocytes, eosinophils, basophils, and monocytes) at Weeks 4, 12, and 16 | Baseline, Weeks 4, 12, and 16
  Platelets, leukocytes, neutrophils, lymphocytes, eosinophils, basophils, and monocytes will be measured in number of blood cells per liter (10^9/L)
Mean Change from Baseline in Hematology Laboratory Analyses (erythrocytes) | Baseline, Week 4, 12, and 16
  Erythrocytes will be measured in number of red blood cells per liter (10^12/L).
Incidence rate for Positive, Negative, Missing Plasma Anti-Bimekizumab Antibodies at Baseline and Week 16 | Baseline and Week 16
  Positive, negative, and missing plasma anti-bimekizumab antibodies detection prior to and following IMP administration during the Initial Treatment Period.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (16):
- United States (10):
  - Hs0006 50175, Phoenix, Arizona
  - Hs0006 50708, Roseville, California
  - Hs0006 50199, Miami, Florida
  - Hs0006 50178, Clarkston, Michigan
  - Hs0006 50710, Fort Gratiot, Michigan
  - Hs0006 50711, Troy, Michigan
  - Hs0006 50712, Brooklyn, New York
  - Hs0006 50706, Chapel Hill, North Carolina
  - Hs0006 50202, Fairborn, Ohio
  - Hs0006 50201, Arlington, Texas
- Germany (2):
  - Hs0006 40326, Berlin
  - Hs0006 40747, Mainz
- Poland (4):
  - Hs0006 40625, Lodz
  - Hs0006 40761, Warsaw
  - Hs0006 40095, Wroclaw
  - Hs0006 40845, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org